CLINICAL TRIAL: NCT05138055
Title: The NOrwegian Tick-borne Encephalitis Study - NOTES: An Observational Study on Clinical Features, Long-term Outcomes and Immune Characteristics
Brief Title: The NOrwegian Tick-borne Encephalitis Study
Acronym: NOTES
Status: Active, not recruiting | Type: Observational
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: Sykehuset i Vestfold HF (Other); Norwegian Institute of Public Health (Other Government); Sorlandet Hospital HF (Other Government); Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 96505
Record Dates: First submitted 2021-02-03; First posted 2021-11-30 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Tick-Borne Encephalitis, European
MeSH Terms: conditions — Encephalitis, Tick-Borne

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and csf
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
During 2018, 2019, and 2020, the reported TBE-cases have increased markedly in Norway. Surveillance studies conducted by the Norwegian Institute of Public Health demonstrate that cases are associated with tick bites in the coastal areas of the Agder, Buskerud, and Vestfold and Telemark counties There is a urgent need for more knowledge of the consequences of TBE in Norway, in particular the identification of patients at risk of long-term sequela. Hence, the overall objective of this project is to gain more knowledge about the natural course of TBE in Norway, and its impact on long-term health-related quality of life and associated factors. Clinical data, biological sampling and PROMs are collected from TBE-infected patients admitted to three hospitals within the epidemic region in Norway.

DETAILED DESCRIPTION:
This project is designed as a multicenter study divided into four sub-studies:

Substudy 1: A retrospective descriptive study of the clinical features and objective findings of the acute phase of the TBE-patients diagnosed with TBE in South-East Norway during 2018, 2019 and 2020.

Substudy 2: A prospective multicenter study of health related QOL one year after hospitalization with TBE in South-East Norway from 2019 - 2023. The self-reported health-related QOL (assesedby SF-36) of the TBE-patients will be compared with the SF-36 reference values in the Norwegian population.

Substudy 3: A prospective multicenter study of self-reported cognitive function one year after hospitalization with TBE in South-East Norway from 2019- 2023. The cognitive function, measured by PROMS, will be compared with PROMS from an included reference group from the patient's social environment.

Substudy 4: Analyses of biological samples collected at baseline, 3 months and 12 months after hospitalization for TBE in patients included in substudy 2 and 3. These analyses will be conducted to gain more knowledge of the pathogenesis of TBE infection and in particular, which molecular pathways and biomarkers that characterize the TBE infected patients who are hospitalized in Norway. Analyses to identify associations between the acute inflammatory response and long-term outcome will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient: The patients diagnosed with acute infection with TBEV at admission.
2. Control: same age (plus/minus 4 years), level of education (plus minus 2 years) and the same gender as patient.

Exclusion Criteria:

1. Patient: Patients who turn out to have different diagnose than acute infections with TBEV.
2. Control: Previously infection with tick-borne encephalitis virus.
3. The patients who were diagnosed with typical symptoms and only TBEV IgM-test must take a blood sample for IgG analyses. If the TBE IgG analysis is negative, the patient will be excluded.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Study population in substudy 1. Patients > 16 years old diagnosed with acute infection caused by TBEV. The hospitals involved are Telemark and Vestfold. Study population in substudy 2. Patients > 16 years old diagnosed with acute infection caused by TBEV. The hospitals involved are Telemark, Vestfold and Sørlandet.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To describe the acute phase clinical and immunological characteristics of TBE in Norway | 4 years
  clinical features and objective findings of the acute phase of the TBE-patients diagnosed with TBE in South-East Norway during 2018-2021
To investigate the impact of TBEV infection on health-related QOL in a one year follow-up study of a Norwegian patient cohort | 4 years
  A prospective multicenter study of health-related QOL one year after hospitalization with TBE in South-East Norway from 2019-2022. The self-reported health-related QOL (assessed by SF-36) of the TBE-patients, will be compared with the SF-36 reference values in the Norwegian population.
To investigate the impact of TBEV infection on long-term cognitive function in a one year follow-up study of a Norwegian patient cohort | 5 years
  A prospective multicenter study of self-reported cognitive function by BRIEF, FSS, HADS and EMQ, one year after hospitalization with TBE in South-East Norway from 2019-2022. The cognitive function, measured by PROMS, will be compared with PROMS from an included reference group from the patient's social environment.
To identify biomarkers in the cerebrospinal fluid (CSF) and blood, which serve as predictors for TBE severity and long-term complaints | 5 years
  FS-36 and BRIEF

CONTACTS AND LOCATIONS:
Overall Officials: Hege Kersten, PhD, Study Director — Study director
Locations (3):
- Norway (3):
  - Sykehuset Telemark HF, Skien, Telemark
  - Sykehuset Sørlandet HF, Arendal
  - Sykehuset i Vestfold, Tønsberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Veje M, Nolskog P, Petzold M, Bergstrom T, Linden T, Peker Y, Studahl M. Tick-Borne Encephalitis sequelae at long-term follow-up: a self-reported case-control study. Acta Neurol Scand. 2016 Dec;134(6):434-441. doi: 10.1111/ane.12561. Epub 2016 Jan 26. PMID 26810689